CLINICAL TRIAL: NCT06224049
Title: A Clinical Study to Evaluate the Safety, Tolerability and Initial Efficacy of Targeted Haploidentical Neoantigen T Cell Injection (hNeo-T) in the Treatment of Relapsed or Refractory EBV-positive T-cell Lymphoma
Brief Title: Treatment of Relapsed or Refractory Epstein-Barr Virus Positive T-cell Lymphoma With hNeo-T
Acronym: GI-hNeoT-01
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: BGI, China (Other)
Collaborators: Shenzhen University General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGI-006; KYLLHS-20230102C (Other: Ethics Committee of Shenzhen University General Hospital)
Record Dates: First submitted 2023-11-13; First posted 2024-01-25 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: T-cell Lymphoma
Keywords: T-cell lymphomas; Epstein-Barr Virus; hNeo-T
MeSH Terms: conditions — Lymphoma, T-Cell; Epstein-Barr Virus Infections | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- hNeo-T (Experimental): The escalating doses of hNeo-T in this study will be 5*10^7 cells and1*10^8 cells.
  Interventions: Biological: hNeo-T; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Biological: hNeo-T — After subject screening, peripheral blood mononuclear cell （PBMC） donors matching half or more of the subject's HLA matching will undergo blood collection to prepare hNeo-T. hNeo-T preparation is expected to be 25-30 days after blood collection. In this study, the bridging therapy will be allowed before Chemotherapy preconditioning, and the investigators will decide whether to use it. Chemotherapy preconditioning will be performed before hNeo-T transfusion. If the absolute value of lymphocyte (LYM) before pretreatment is <0.8×10^9/L and the subject meets the criteria for cell transfusion, the chemotherapy preconditioning will not be performed and subsequent cell transfusion can be performed directly.
Drug: Cyclophosphamide — Chemotherapy preconditioning will be performed before hNeo-T transfusion.
Drug: Fludarabine — Chemotherapy preconditioning will be performed before hNeo-T transfusion

SUMMARY:
Objective: To evaluate the safety and tolerability of hNeo-T injection in patients with relapsed or refractory EBV-positive T-cell lymphoma.

Secondary objective: To evaluate the effectiveness of hNeo-T injection, and to evaluate the objective response rate (ORR) and disease control rate (DCR) by Lugano2014 criteria; Progression-free survival (PFS), duration of response (DOR), and overall survival (OS ) followed.

Objective of the exploratory study: To investigate the in vivo process of hNeo-T injection and describe the activity and related biological functions of hNeo-T cells in vivo, including but not limited to.

DETAILED DESCRIPTION:
This is a single arm,open label and non-randomized clinical trial with a planned enrollment of 6-12 participants to evaluate the safety and tolerability of hNeo-T injection, determine dose-limiting toxicity (DLT), explore the maximum tolerated dose (MTD), or the recommended dosage for later clinical studies.

The DLT observation period is 28 days after the infusion of hNeo-T injection. In the first stage, 3 subjects will be enrolled in the experiment of the first dose group (total number of cells is 5×10^7/ bag). If DLT does not appear during the experiment, the study will enter the second stage after safety assessment and analysis, and 3 subjects will be enrolled in the experiment of the second dose group (total number of cells is 1×10^8/ bag) in this stage.

If DLT occurs in one of the 3 subjects , three more subjects will be added to the dose group. If no additional DLT occurs, the study will enter the next dose group; If additional DLT occurs, enrollment in the group will be stopped and the dose will be defined as an intolerable dose; If DLT occurs in two or more of the 3 subjects, enrollment in the dose group will be discontinued and the dose will be defined as an intolerable dose;

After climbing to an intolerable dose, there will be a discussion to decide whether to explore an intermediate dose or to define the dose level as MTD; If MTD is not defined in the high-dose group, the high-dose group will be used as the final climbing dose. If a higher dose will be planned, a follow-up clinical study can only be carried out after evaluation,discussion and consensus.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, and ≤75 years old, gender is not limited;
2. Must have histologically or cytologically confirmed T-cell lymphoma with at least one measurable tumor lesion (according to Lugano2014 criteria);
3. The subject's HLA type is HLA-A0201/1101/2402/0203 (containing at least one of the subtypes, as determined by the test report issued by the central laboratory), and there is at least one healthy donor who is a semi-matching HLA type or more with the subject. At least one of the HLA matching loci is HLA-A0201/1101/2402/0203；
4. The subject has been previously determined to be EBV positive or has been determined to be EBV positive after testing;
5. The subject has paraffin-embedded tumor tissue/section or biopsy tumor tissue within 2.5 years (tissue biopsy is recommended for subjects with easy-to-sample tumor lesions and consent to biopsy), and these tissues are qualified by gene sequencing data. And the tumor neoantigen screening qualified;
6. Disease progression after adequate first-line systemic treatment, or disease progression ≥2 cycles (PD) after first-line or above systemic systemic treatment, or ≥4 cycles without remission (CR or PR). Remarks: The first-line systemic treatment should refer to the latest version of the "Lymphoma Diagnosis and Treatment Guide" issued by China's "Chinese Society of Clinical Oncology".
7. Volunteer to participate in clinical studies; I or legal guardian fully understand and know the study and sign the informed consent; Willing to follow and be able to complete all test procedures;
8. ECOG score ≤1 score;
9. Have venous access to meet venous blood collection;
10. The survival time is expected to be ≥6 months;
11. The subjects are willing to use a reliable method of contraception during treatment and within 3 months after the end of treatment, and the blood pregnancy test of women of childbearing age is negative;
12. Laboratory test results and vital organ functions meet the following requirements: 1) *HIV antibody negative; No active syphilis infection; Negative antibodies to hepatitis C virus; HBV DNA detection value is lower than the upper limit of normal value; 2) Blood routine: absolute value of neutrophil (ANC) ≥1×10^9/L, platelet count (PLT) ≥75×10^9/L, hemoglobin concentration (HGB) ≥80g/L; 3) Blood biochemistry: glutamic-pyruvic transaminase (ALT) and glutamic-oxalic transaminase (AST) ≤3 times the upper limit of normal (ULN) (ALT and AST≤5 times ULN in liver metastasis subjects); Serum creatinine ≤1.5 ULN; Total bilirubin ≤1.5 ULN, or total bilirubin <3 ULN for subjects with GilbertsSyndrome; 4) Coagulation function: prothrombin time (PT) and International standard ratio (INR) ≤1.5 times ULN, activated partial thromboplastin time (APTT) ≤1.5 times ULN (for subjects taking anticoagulant drugs for a long time, the coagulation related indexes can meet the normal value range after medication); 5) Left ventricular ejection fraction (LVEF) ≥50%;
13. Before administration with Chemotherapy preconditioning: 1) Any chemotherapy, targeted drugs, immune checkpoint inhibitors, other drugs studied in clinical trials, Chinese medicines with anti-tumor indications, and other anti-tumor treatments received have passed the 4-week washout period, and the toxic side effects have returned to grade 1 or lower (excluding hair loss, vitiligo, and other events that the investigator has judged to be tolerated); 2) If major surgery is performed within 3 weeks, adverse reactions have recovered to grade 1 or lower.

Exclusion Criteria:

1. Pregnant or lactating women;
2. People with a history of severe hypersensitivity to the cells used in this study and to any drugs;
3. Patients with a history of organ transplantation, excluding hematopoietic stem cell transplantation;
4. History of allogeneic hematopoietic stem cell transplantation; Acute or chronic graft-versus-host disease (GVHD);
5. Clear central nervous system involvement of lymphoma, including parenchyma, meningeal invasion or spinal cord compression;
6. Any person with active autoimmune disease or who has a history of autoimmune disease that the investigator has determined to be ineligible for this study, including but not limited to the following diseases: Such as systemic lupus erythematosus, immune-related neuropathy, multiple sclerosis, Guillain-Barre syndrome, myasthenia gravis, connective tissue diseases, inflammatory bowel diseases including Crohn's disease and ulcerative colitis (except for patients with vitiligo, eczema, type I diabetes, rheumatoid arthritis and other joint diseases, sjogren's syndrome and psoriasis controlled with topical drugs);
7. Uncontrolled concomitant or infectious diseases, such as acutely active infected persons requiring systemic antibiotic, antiviral or antifungal treatment within 2 weeks prior to enrollment;
8. Severe impairment of liver or kidney function (liver or kidney therapy but not controllable, biochemical indicators are not yet able to meet the criteria for inclusion in Article 11), or uncontrolled diabetes, pulmonary fibrosis, interstitial lung disease, acute lung disease, or medically poorly controlled hypertension (systolic blood pressure >160mmHg and/or diastolic blood pressure >90mmHg), Or cardiovascular and cerebrovascular diseases of clinical significance (e.g. active), For example, cerebrovascular accident (within 6 months before the signing of the informed consent), myocardial infarction (within 6 months before the signing of the informed consent), unstable angina, congestive heart failure classified by the New York Heart Association (NYHA) as class II or above, severe arrhythmia that cannot be controlled with drugs, and electrocardiogram results showing clinical significance in 3 consecutive times (each interval of at least 5 minutes) The presence of abnormalities determined by the investigator to affect subsequent cell therapy, or mental illness and substance abuse, or any condition that the investigator believes may increase the risk of the subject or interfere with the test results;
9. Subjects who were scheduled to receive glucocorticoids (prednisone or equivalent dose >10mg/ day) or other immunosuppressants for a condition within 2 weeks prior to lymphocyte clearance preconditioning administration and during the study period were excluded. Remarks: In the absence of active autoimmune disease, prednisone or an equivalent adrenal drug dose ≤10mg/ day is allowed to substitute administration; Subjects were allowed to use topical, ocular, intraarticular, intranasal, and inhaled corticosteroids (with very low systemic absorption);
10. Subject is scheduled to receive immunomodulatory drugs (such as interferon, GM-CSF, thymosin, gamma globulin, etc.) within 2 weeks before lymphocyte clearance preconditioning administration and during the study period due to certain conditions;
11. The investigator evaluates that the subject is unable or unwilling to comply with the requirements of the study protocol;
12. Those with functional defects of genes related to antigen presentation, antigen recognition and cell killing detected by sequencing;
13. History of other malignant tumors within the past 5 years; Excluding curable basal or squamous cell skin cancer, superficial bladder or prostate carcinoma in situ, cervical carcinoma in situ or breast carcinoma in situ;
14. The subject has any disease or medical condition that may affect the evaluation of the safety or efficacy of the investigational drug.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety assessment (Evaluation of treatment-related adverse events according to CTCAEv5.0) | The first dose will be administered until 28 days after the last dose
  To determine the incidence of AE and SAE in clinical trials

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 48 weeks
  The total number of subjects with complete response (CR) and partial response (PR) confirmed according to Lugano2014 criteria (i.e., CR+PR) and the proportion of subjects in the corresponding analysis set
Disease control rate (DCR) | Up to 48 weeks
  The total number of subjects with CR, PR, and stable disease (SD) confirmed according to Lugano2014 criteria (i.e. CR+PR+SD) and the proportion of subjects in the corresponding analysis set
Progression free survival (PFS) | Up to 52 weeks
  According to the Lugano2014 criteria, the time between the start of cell transfusion and the first recorded date of disease progression (PD) or death. If no disease progression is observed, the deletion date should be the date of the last tumor measurement, and if there is no baseline and/or tumor evaluation after transfusion, the PFS will be deleted to the cell transfusion date. Detailed rules on deletion will be described in the statistical analysis plan.
Duration of response (DOR) | Up to 36 weeks
  According to the Lugano2014 criteria, the time between a subject's first identification with CR or PR and the first recording of PD or the date of death, depending on which occurs first. For subjects who do not experience disease progression after a combined response, the duration of response will be deleted at the last evaluable tumor measurement date.
Overall survival (OS) | Up to 72 weeks
  The time from cell transfusion to death who have completed the prescribed dose. If the subjects is lost to follow-up, the last known date of survival will be OS deletion time.

CONTACTS AND LOCATIONS:
Overall Officials: LiXin Wang, Doctor, Principal Investigator — Shenzhen University General Hospital
Locations (1):
- ShenZhen University General Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Comoli P, Basso S, Riva G, Barozzi P, Guido I, Gurrado A, Quartuccio G, Rubert L, Lagreca I, Vallerini D, Forghieri F, Morselli M, Bresciani P, Cuoghi A, Paolini A, Colaci E, Marasca R, Cuneo A, Iughetti L, Trenti T, Narni F, Foa R, Zecca M, Luppi M, Potenza L. BCR-ABL-specific T-cell therapy in Ph+ ALL patients on tyrosine-kinase inhibitors. Blood. 2017 Feb 2;129(5):582-586. doi: 10.1182/blood-2016-07-731091. Epub 2016 Dec 7. PMID 27927646
- [Background] Chen Y, Zhao H, Luo J, Liao Y, Dan X, Hu G, Gu W. A phase I dose-escalation study of neoantigen-activated haploidentical T cell therapy for the treatment of relapsed or refractory peripheral T-cell lymphoma. Front Oncol. 2022 Nov 10;12:944511. doi: 10.3389/fonc.2022.944511. eCollection 2022. PMID 36439517
- [Background] Zacharakis N, Chinnasamy H, Black M, Xu H, Lu YC, Zheng Z, Pasetto A, Langhan M, Shelton T, Prickett T, Gartner J, Jia L, Trebska-McGowan K, Somerville RP, Robbins PF, Rosenberg SA, Goff SL, Feldman SA. Immune recognition of somatic mutations leading to complete durable regression in metastatic breast cancer. Nat Med. 2018 Jun;24(6):724-730. doi: 10.1038/s41591-018-0040-8. Epub 2018 Jun 4. PMID 29867227
- [Background] Keskin DB, Anandappa AJ, Sun J, Tirosh I, Mathewson ND, Li S, Oliveira G, Giobbie-Hurder A, Felt K, Gjini E, Shukla SA, Hu Z, Li L, Le PM, Allesoe RL, Richman AR, Kowalczyk MS, Abdelrahman S, Geduldig JE, Charbonneau S, Pelton K, Iorgulescu JB, Elagina L, Zhang W, Olive O, McCluskey C, Olsen LR, Stevens J, Lane WJ, Salazar AM, Daley H, Wen PY, Chiocca EA, Harden M, Lennon NJ, Gabriel S, Getz G, Lander ES, Regev A, Ritz J, Neuberg D, Rodig SJ, Ligon KL, Suva ML, Wucherpfennig KW, Hacohen N, Fritsch EF, Livak KJ, Ott PA, Wu CJ, Reardon DA. Neoantigen vaccine generates intratumoral T cell responses in phase Ib glioblastoma trial. Nature. 2019 Jan;565(7738):234-239. doi: 10.1038/s41586-018-0792-9. Epub 2018 Dec 19. PMID 30568305
- [Background] Hilf N, Kuttruff-Coqui S, Frenzel K, Bukur V, Stevanovic S, Gouttefangeas C, Platten M, Tabatabai G, Dutoit V, van der Burg SH, Thor Straten P, Martinez-Ricarte F, Ponsati B, Okada H, Lassen U, Admon A, Ottensmeier CH, Ulges A, Kreiter S, von Deimling A, Skardelly M, Migliorini D, Kroep JR, Idorn M, Rodon J, Piro J, Poulsen HS, Shraibman B, McCann K, Mendrzyk R, Lower M, Stieglbauer M, Britten CM, Capper D, Welters MJP, Sahuquillo J, Kiesel K, Derhovanessian E, Rusch E, Bunse L, Song C, Heesch S, Wagner C, Kemmer-Bruck A, Ludwig J, Castle JC, Schoor O, Tadmor AD, Green E, Fritsche J, Meyer M, Pawlowski N, Dorner S, Hoffgaard F, Rossler B, Maurer D, Weinschenk T, Reinhardt C, Huber C, Rammensee HG, Singh-Jasuja H, Sahin U, Dietrich PY, Wick W. Actively personalized vaccination trial for newly diagnosed glioblastoma. Nature. 2019 Jan;565(7738):240-245. doi: 10.1038/s41586-018-0810-y. Epub 2018 Dec 19. PMID 30568303